CLINICAL TRIAL: NCT04008394
Title: Efficacy and Safety of Anti-CD30 CAR-T Therapy in Patients With Refractory/Relapsed Lymphocyte Malignancies：a Single-center, Open, Single-arm Clinical Study.
Brief Title: Anti-CD30 CAR-T Therapy in Patients With Refractory/Relapsed Lymphocyte Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Bio-Raid Biotechnology Co, Ltd. China (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHUH-CART-CD30-01
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Adult T-Cell Lymphoma/Leukaemia; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; NK/T-cell Lymphoma; Peripheral T Cell Lymphoma; Hodgkin Lymphoma
Keywords: CD-30 CART; Refractory/Relapsed; lymphocyte malignancies
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell, Peripheral; Hodgkin Disease; Recurrence

STUDY DESIGN:
Intervention Model Description: Single-center,Open,One-arm Clinical Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD30 CAR T cells (Experimental): Patients receive CD30 CAR-T cells transduced with a lentiviral vector on day 0 in the absence of disease progression or unacceptable toxicity. Autologous 3th generation anti-CD30 CAR T cells.
  Interventions: Genetic: Anti-CD30 CAR T cells

INTERVENTIONS:
Genetic: Anti-CD30 CAR T cells — Patients receive CD30 CAR-T cells transduced with a lentiviral vector on day 0 in the absence of disease progression or unacceptable toxicity. Autologous 3th generation anti-CD30 CAR T cells.

SUMMARY:
The overall purpose of this study is to explore the safety and therapeutic effect of CD30-targeted chimeric antigen receptor T(CAR-T) cells in the treatment of Refractory/Relapsed lymphocyte malignancies.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells (CAR-T cells) have the capabilities to recognize tumor associated antigen and kill tumor cells specifically. CD30 is originally described as a marker of Hodgkin's and R-S cells in Hodgkin's lymphoma. CD30 antibody has been applied to treat lymphocyte derived malignancies. To explore the potency of CD30 in CAR-T therapy, this trial is designed and conducted to test the safety and efficacy of CD30-targeted CAR-T in Refractory/Relapsed lymphocyte malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.
2. Male or female patients aged 18 to 70 years (including 18 and 70 years old).
3. Pathological and histological examination confirmed CD30+ lymphocyte malignancies, and patients currently have no effective treatment options, such as chemotherapy or recurrence after hematopoietic stem cell transplantation; or patients voluntarily choose Anti-CD30 CAR-T as rescue treatment.
4. CD30+ lymphocyte malignancies:

   1. Adult T-cell leukemia/lymphoma
   2. Anaplastic large cell lymphoma (ALCL);
   3. Angioimmunoblastic T-cell Lymphoma (AITL);
   4. NK/T-cell lymphoma;
   5. Peripheral T-cell lymphoma (PTCL);
   6. Hodgkin lymphoma;
5. Subjects:

   1. There are still residual lesions after major treatment, and they are not suitable for HSCT (auto/allo-HSCT);
   2. Recurrence occurs after CR1, and HSCT (auto/allo-HSCT) is not selected or suitable because of self-willingness;
   3. After hematopoietic stem cell transplantation or cellular immunotherapy, the patient suffered relapse or did not remission.
6. Having a measurable or evaluable lesion.
7. Patient's main organs function well：

   1. Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and
   2. total bilirubin≤34.2μmol/L
   3. Renal function: Creatinine < 220μmol/L.
   4. Pulmonary function: Indoor oxygen saturation≥95%.
   5. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥40%.
8. The patients did not receive any anticancer treatments such as chemotherapy, radiotherapy and immunotherapy (such as immunosuppressive drugs) within 4 weeks before admission, and the toxicity related to previous treatments had returned to < 1 level at admission (except for low toxicity such as alopecia).
9. The patient's peripheral superficial venous blood flow smoothly, which can meet the needs of intravenous drip.
10. Patient ECOG score≤2, Estimated survival time≥3 months.

Exclusion Criteria:

1. Women who are pregnant (urine/blood pregnancy test positive) or lactating.
2. Male or female with a conception plan in the past 1 years.
3. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 years after enrollment.
4. Uncontrolled infectious disease within 4 weeks prior to enrollment.
5. Active hepatitis B/C virus.
6. HIV infected patients.
7. Suffering from a serious autoimmune disease or immunodeficiency disease.
8. The patient is allergic and is allergic to macromolecular biopharmaceuticals such as antibodies or cytokines.
9. The patient participated in other clinical trials within 6 weeks prior to enrollment.
10. Systemic use of hormones within 4 weeks prior to enrollment (except for patients with inhaled corticosteroids).
11. Have a history of epilepsy or other central nervous system diseases.
12. Having drug abuse/addiction.
13. According to the researcher's judgment, the patient has other unsuitable grouping conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 3 years
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0).

SECONDARY OUTCOMES:
One-month remission rate | 1 month
  Response to CAR-T therapy was assessed on day 30 (±2), against the National Comprehensive Cancer Network (NCCN, Version 1.2015).
Overall survival | 3 years
  OS was calculated from the first CAR-T cell infusion to death or last follow-up (censored).
Event-free survival | 3 years
  EFS was calculated from the first CAR-T cell infusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit (censored).
Relapse-free survival | 3 years
  RFS was calculated from the first CAR-T cell infusion to relapse or last visit (censored).
Quantity of anti-CD30 CAR-T cells in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) quantity of CAR-T cells were determined by means of flow cytometry.
Quantity of anti-CD30 CAR copies in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) quantity of anti-CD30 CAR copies were determined by means of qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D. Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No